CLINICAL TRIAL: NCT00002633
Title: Phase III Randomized Trial Comparing Total Androgen Blockade Versus Total Androgen Blockade Plus Pelvic Irradiation in Clinical Stage T3-4, N0, M0 Adenocarcinoma of the Prostate
Brief Title: Hormone Therapy With or Without Surgery or Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network); Medical Research Council (Other Government)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR3; CAN-NCIC-PR3 (Registry Identifier: NCI US PDQ); ECOG-JPR03 (Other: ECOG); MRC-PR07 (Other: MRC); SWOG-JPR3 (Other: SWOG); EU-99013 (Other: EU); NCI-T94-0110O (Other Grant/Funding Number: NCI); ISRCTN24991896 (Registry Identifier: ISRCTN); CDR0000064065 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Buserelin; Flutamide; Goserelin; Leuprolide; nilutamide; Orchiectomy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total Androgen Blockade (Active Comparator)
  Interventions: Drug: bicalutamide; Drug: buserelin; Drug: flutamide; Drug: goserelin; Drug: leuprolide acetate; Drug: nilutamide; Procedure: orchiectomy
- Total Androgen Blockade Vs TA Blockade Plus Pelvic Irradiation (Active Comparator)
  Interventions: Drug: bicalutamide; Drug: buserelin; Drug: flutamide; Drug: goserelin; Drug: leuprolide acetate; Drug: nilutamide; Procedure: orchiectomy; Radiation: radiation therapy

INTERVENTIONS:
Drug: bicalutamide — Antiandrogen (optional with orchiectomy) Flutamide 250 mg po TID or Nilutamide 100 mg po TID x 1 mo; then 150 mg po QD or Bicalutamide 50 mg po QD PLUS (patient's choice) Bilateral orchiectomy or LHRH agonist Goserelin 3.6 mg SC (abd) q28d or 10.8 mg SC (abd) Q3mos or Leuprolide 7.5 mg IM q28d (Leuprorelin 3.75 mg) or 22.5 mg IM Q3mos (Leuprorelin 11.25 mg) or 30 mg IM Q4mos or Buserelin 6.3mg SC (abd) Q8wk or 9.45mg SC (abd) Q12wk
Drug: buserelin — Antiandrogen (optional with orchiectomy) Flutamide 250 mg po TID or Nilutamide 100 mg po TID x 1 mo; then 150 mg po QD or Bicalutamide 50 mg po QD PLUS (patient's choice) Bilateral orchiectomy or LHRH agonist Goserelin 3.6 mg SC (abd) q28d or 10.8 mg SC (abd) Q3mos or Leuprolide 7.5 mg IM q28d (Leuprorelin 3.75 mg) or 22.5 mg IM Q3mos (Leuprorelin 11.25 mg) or 30 mg IM Q4mos or Buserelin 6.3mg SC (abd) Q8wk or 9.45mg SC (abd) Q12wk
Drug: flutamide — Antiandrogen (optional with orchiectomy) Flutamide 250 mg po TID or Nilutamide 100 mg po TID x 1 mo; then 150 mg po QD or Bicalutamide 50 mg po QD PLUS (patient's choice) Bilateral orchiectomy or LHRH agonist Goserelin 3.6 mg SC (abd) q28d or 10.8 mg SC (abd) Q3mos or Leuprolide 7.5 mg IM q28d (Leuprorelin 3.75 mg) or 22.5 mg IM Q3mos (Leuprorelin 11.25 mg) or 30 mg IM Q4mos or Buserelin 6.3mg SC (abd) Q8wk or 9.45mg SC (abd) Q12wk
Drug: goserelin — Antiandrogen (optional with orchiectomy) Flutamide 250 mg po TID or Nilutamide 100 mg po TID x 1 mo; then 150 mg po QD or Bicalutamide 50 mg po QD PLUS (patient's choice) Bilateral orchiectomy or LHRH agonist Goserelin 3.6 mg SC (abd) q28d or 10.8 mg SC (abd) Q3mos or Leuprolide 7.5 mg IM q28d (Leuprorelin 3.75 mg) or 22.5 mg IM Q3mos (Leuprorelin 11.25 mg) or 30 mg IM Q4mos or Buserelin 6.3mg SC (abd) Q8wk or 9.45mg SC (abd) Q12wk
Drug: leuprolide acetate — Antiandrogen (optional with orchiectomy) Flutamide 250 mg po TID or Nilutamide 100 mg po TID x 1 mo; then 150 mg po QD or Bicalutamide 50 mg po QD PLUS (patient's choice) Bilateral orchiectomy or LHRH agonist Goserelin 3.6 mg SC (abd) q28d or 10.8 mg SC (abd) Q3mos or Leuprolide 7.5 mg IM q28d (Leuprorelin 3.75 mg) or 22.5 mg IM Q3mos (Leuprorelin 11.25 mg) or 30 mg IM Q4mos or Buserelin 6.3mg SC (abd) Q8wk or 9.45mg SC (abd) Q12wk
Drug: nilutamide — Antiandrogen (optional with orchiectomy) Flutamide 250 mg po TID or Nilutamide 100 mg po TID x 1 mo; then 150 mg po QD or Bicalutamide 50 mg po QD PLUS (patient's choice) Bilateral orchiectomy or LHRH agonist Goserelin 3.6 mg SC (abd) q28d or 10.8 mg SC (abd) Q3mos or Leuprolide 7.5 mg IM q28d (Leuprorelin 3.75 mg) or 22.5 mg IM Q3mos (Leuprorelin 11.25 mg) or 30 mg IM Q4mos or Buserelin 6.3mg SC (abd) Q8wk or 9.45mg SC (abd) Q12wk
Procedure: orchiectomy — Optional orchiectomy
Radiation: radiation therapy — Radical Radiation Therapy - (65-69 Gy; 35-37 treatments)
  Arms: Total Androgen Blockade Vs TA Blockade Plus Pelvic Irradiation

SUMMARY:
RATIONALE: Hormones can stimulate the growth of prostate cancer cells. Hormone therapy may fight prostate cancer by reducing the production of androgens. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether hormone therapy plus surgery is more effective than hormone therapy plus radiation therapy for prostate cancer.

PURPOSE: This randomized phase III trial is studying giving hormone therapy alone to see how well it works compared to giving hormone therapy together with bilateral orchiectomy or radiation therapy in treating patients with stage III or stage IV prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival, disease specific survival, and time to progression in patients with locally advanced adenocarcinoma of the prostate treated with total androgen suppression with or without pelvic irradiation.
* Compare the symptomatic control as measured by the rates of surgical interventions needed for control of local disease (e.g., transurethral resections, stent insertions, nephrostomies, and colostomies) in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare the sensitivity of the EORTC-QLQ-C30+3 and a trial-specific checklist (PR17) with the FACT-P questionnaire in measuring changes in quality of life of patients treated with these regimens.

OUTLINE: This a randomized, multicenter study. Patients are stratified according to center, initial PSA level (less than 20 vs 20-50 vs greater than 50 ng/mL), method of node staging (clinical [no CT scan] vs radiological [CT scan negative] vs surgical), Gleason score (less than 8 vs 8-10), prior hormonal therapy (excluding orchiectomy) (yes vs no), and choice of hormonal therapy (bilateral orchiectomy with or without antiandrogen vs luteinizing hormone-releasing hormone [LHRH] with antiandrogen). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive antiandrogen therapy comprising oral flutamide every 8 hours, oral nilutamide every 8 hours for 1 month and then once daily, or oral bicalutamide once daily. Patients also choose to undergo bilateral orchiectomy or LHRH agonist therapy comprising goserelin subcutaneously (SC) every 4 weeks (short-acting formulation) or every 3 months (long-acting formulation), leuprolide intramuscularly every 4 weeks (short-acting formulation) or every 3 months (long-acting formulation), or buserelin SC every 8 weeks or every 12 weeks. Patients choosing orchiectomy may receive an antiandrogen for at least 6 weeks before surgery to counter any flare phenomenon and may continue the antiandrogen after surgery (at the physician's discretion).
* Arm II: Patients undergo total androgen ablation as in arm I. Patients with node-negative dissection undergo radiotherapy 5 days a week for 6.5-7 weeks. All other patients undergo radiotherapy 5 days a week for 5 weeks, followed by boost radiotherapy 5 days a week for 2-2.4 weeks.

Hormonal therapy on both arms continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, on the last day of radiotherapy, at 6 months, and then every 6 months thereafter.

Patients are followed at 1, 2, and 6 months and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 1,200 patients will be accrued for this study within 7.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven locally advanced adenocarcinoma of the prostate, defined as 1 of the following:

  * T3-4, N0 or NX, M0
  * T2, PSA greater than 40 µg/L
  * T2, PSA greater than 20 µg/L AND Gleason score at least 8
* Diagnosis made within the past 6 months
* Gleason score and PSA known
* Pelvic lymph nodes must be clinically negative

  * Lymph nodes no more than 1.5 cm in greatest diameter by CT scan or MRI of the pelvis
  * Negative needle aspirate required for any lymph node more than 1.5 cm
  * If a lymph node dissection was performed, it must be histologically negative
* No small cell or transitional cell carcinoma by biopsy
* No bony metastases by bone scan

PATIENT CHARACTERISTICS:

Age:

* Under 80

Performance status:

* ECOG 0-2

Life expectancy:

* At least 5 years excluding malignancy

Hematopoietic:

* Hemoglobin at least 10.0 g/dL
* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2 times upper limit of normal (ULN)
* SGOT and SGPT less than 2 times ULN
* Alkaline phosphatase less than 2 times ULN
* No history of chronic liver disease

Renal:

* Creatinine less than 2 times ULN

Other:

* No contraindication to wide-field pelvic irradiation (e.g., inflammatory bowel disease or severe bladder irritability)
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Prior hormonal therapy within the past 12 weeks allowed provided the following conditions are met:

  * Negative bone scan before beginning any hormonal therapy
  * Extracapsular extension remains palpable on rectal re-exam
  * Baseline PSA known before beginning any hormonal therapy
* At least 4-6 weeks since prior 5-alpha-reductase inhibitor (e.g., finasteride) for benign prostatic hypertrophy

Radiotherapy:

* No prior pelvic irradiation

Surgery:

* No prior radical prostatectomy
* Prior transurethral resection of the prostate allowed

Other:

* No prior cytotoxic anticancer therapy
* No other prior treatment for prostate cancer
* No other concurrent anticancer therapy unless documented disease progression

Max Age: 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 1995-02-08 (Actual); Primary Completion 2011-09-23 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 10 years

SECONDARY OUTCOMES:
Disease specific survival | 10 years
Time to disease progression | 10 years
Symptomatic local control measured by surgical intervention rate | 10 years
Quality of life assessed by EORTC-QLQ-C30 + 3 and a trial-specific checklist (PR17) or the FACT-P questionnaire | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Padraig R. Warde, MB, MRCPI, FRCPC, Study Chair — Princess Margaret Hospital, Canada; Richard R. Whittington, MD, Study Chair — Abramson Cancer Center at Penn Medicine; Srinivasan Vijayakumar, MD, Study Chair — Michael Reese Hospital and Medical Center; Patricia Lillis-Hearne, MD, Study Chair — Brooke Army Medical Center; Malcolm D. Mason, MD, Study Chair — Velindre NHS Trust
Locations (15):
- Canada (15):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Regional Cancer Program of the Hopital Regional, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Warde P, Mason M, Ding K, Kirkbride P, Brundage M, Cowan R, Gospodarowicz M, Sanders K, Kostashuk E, Swanson G, Barber J, Hiltz A, Parmar MK, Sathya J, Anderson J, Hayter C, Hetherington J, Sydes MR, Parulekar W; NCIC CTG PR.3/MRC UK PR07 investigators. Combined androgen deprivation therapy and radiation therapy for locally advanced prostate cancer: a randomised, phase 3 trial. Lancet. 2011 Dec 17;378(9809):2104-11. doi: 10.1016/S0140-6736(11)61095-7. Epub 2011 Nov 2. PMID 22056152
- [Derived] Brundage M, Sydes MR, Parulekar WR, Warde P, Cowan R, Bezjak A, Kirkbride P, Parliament M, Moynihan C, Bahary JP, Parmar MK, Sanders K, Chen BE, Mason MD. Impact of Radiotherapy When Added to Androgen-Deprivation Therapy for Locally Advanced Prostate Cancer: Long-Term Quality-of-Life Outcomes From the NCIC CTG PR3/MRC PR07 Randomized Trial. J Clin Oncol. 2015 Jul 1;33(19):2151-7. doi: 10.1200/JCO.2014.57.8724. Epub 2015 May 26. PMID 26014295
- [Derived] Mason MD, Parulekar WR, Sydes MR, Brundage M, Kirkbride P, Gospodarowicz M, Cowan R, Kostashuk EC, Anderson J, Swanson G, Parmar MK, Hayter C, Jovic G, Hiltz A, Hetherington J, Sathya J, Barber JB, McKenzie M, El-Sharkawi S, Souhami L, Hardman PD, Chen BE, Warde P. Final Report of the Intergroup Randomized Study of Combined Androgen-Deprivation Therapy Plus Radiotherapy Versus Androgen-Deprivation Therapy Alone in Locally Advanced Prostate Cancer. J Clin Oncol. 2015 Jul 1;33(19):2143-50. doi: 10.1200/JCO.2014.57.7510. Epub 2015 Feb 17. PMID 25691677